CLINICAL TRIAL: NCT07231250
Title: Glofitamab Plus Polatuzumab Vedotin and Zuberitamab in Patients With Newly Diagnosed Diffuse Large B-cell Lymphoma: A Multicenter Phase II Study
Brief Title: Glofitamab Plus Polatuzumab Vedotin and Zuberitamab in Patients With Newly Diagnosed Diffuse Large B-cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li Zhiming (Other)
Responsible Party: Sponsor-Investigator, Li Zhiming, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML45750
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma; Chemo-free Therapy; Bispecific Antibody
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating | interventions — glofitamab; polatuzumab vedotin; Cyclophosphamide; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Trial group (Experimental): After receiving 3 cycles of Glofitamab plus Polatuzumab vedotin and Zuberitamab（Anti-CD20 Monoclonal Antibody）, patients were treated with Glofitamab plus Polatuzumab vedotin and Zuberitamab for 5 cycles if CR or Glofitamab plus Polatuzumab vedotin and Zuberitamab-CHP for 6 cycles if PR/SD based on iPET status.
  Interventions: Drug: Glofitamab; Polatuzumab vedotin; Zuberitamab; Cyclophosphamide; Doxorubicin; Prednisone

INTERVENTIONS:
Drug: Glofitamab; Polatuzumab vedotin; Zuberitamab; Cyclophosphamide; Doxorubicin; Prednisone — Step-up cycle (cycle 1) will comprise intravenous (i.v.) application of obinutuzumab 1,000 mg on D1, followed by i.v. application of polatuzumab vedotin 1.8 mg/kg on D2 and i.v. application of glofitamab in escalating doses of 2.5 mg on D8 and 10 mg on D15.
  Target dose phase (cycle 2-3) will comprise polatuzumab vedotin 1.8 mg/kg, i.v., glofitamab 30 mg i.v. and Zuberitamab 375mg/m2 i.v. on D1 and repeated Q3W.
  Adaptive treatment phase (cycle 4-9) will include two arms with dose cycle guided by PET/CT after C3: i.) If CR, it will comprise polatuzumab vedotin 1.8 mg/kg, i.v.(C4-6) on D1, glofitamab 30 mg i.v. (C4-8) on D2 and Zuberitamab 375mg/m2 i.v. (C4-8) on D1 and repeated Q3W. ii.) if PR or SD, it will comprise polatuzumab vedotin 1.8 mg/kg, i.v .(C4-6) on D1, glofitamab 30 mg i.v. (C4-8) on D8, Zuberitamab-CHP[Zuberitamab 375mg/m2 i.v., cyclophosphamide i.v., doxorubicin i.v., and prednisone p.o. (C4-9)] on D1 and repeated Q3W.

SUMMARY:
This is a multi-center, phase II, prospective study. The main purpose of study is to evaluate the efficacy and safety of Glofitamab plus Polatuzumab vedotin and Zuberitamab in patients with newly diagnosed diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Nearly 1/3 of newly diagnosed DLBCL patients are over 75 years old, with a median age of 66. The number and proportion of patients unable to tolerate conventional immunochemotherapy continue to rise. Serious long-term toxicities associated with chemotherapy (e.g., reproductive effects, secondary malignancies) have created substantial clinical demand for first-line chemotherapy-free regimens. There is an urgent need for more clinical trials to explore the feasibility of chemo-free or chemo-light regimens in previously untreated DLBCL.

The Smart Stop study from MD Anderson is currently exploring chemotherapy-free, response-adapted therapy based on LTRA (Lymphoma Treatment Response Assessment) protocols. Meanwhile, the MOLTO study demonstrated that atezolizumab combined with venetoclax and obinutuzumab provides effective and well-tolerated treatment for previously untreated transformed DLBCL. This evidence above supports chemo-free or chemo-light regimens as a promising new direction for investigation in previously untreated DLBCL.

Early data suggest that Glofit + Pola-R-CHP in 1L DLBCL has promising efficacy and a similar safety profile to Pola-R-CHP and Glofit + R-CHOP.

This is a multi-center, phase II, prospective study. The main purpose of study is to evaluate the efficacy and safety of Glofitamab plus Polatuzumab vedotin and Zuberitamab in patients with newly diagnosed diffuse large B-cell lymphoma. After receiving 3 cycles of Glofitamab plus Polatuzumab vedotin and Zuberitamab（Anti-CD20 Monoclonal Antibody）, patients were treated with Glofitamab plus Polatuzumab vedotin and Zuberitamab for 5 cycles if CR or Glofitamab plus Polatuzumab vedotin and Zuberitamab-CHP for 6 cycles if PR/SD based on iPET status. The primary efficacy endpoint is CR rate at C4D1.

ELIGIBILITY:
Inclusion Criteria:

* The following criteria must be met to be eligible for the study:

  1. Written informed consent.
  2. Age ≥18 years at the time of signing the Informed Consent Form
  3. IPI score 2-5.
  4. ECOG performance status of 0-2.
  5. Histologically confirmed CD20-positive LBCL, including one of the following diagnoses by 2022 WHO classification of lymphoid neoplasms:
* DLBCL, not otherwise specified (NOS) including germinal B-cell type, activated B-cell type
* T-cell/histiocyte-rich large B-cell lymphoma
* Epstein-Barr virus-positive DLBCL, NOS
* Anaplastic lymphoma kinasepositive large B-cell lymphoma
* Kaposi's sarcomaassociated herpesvirus/human herpesvirus-8positive DLBCL
* DLBCL/HGBCL with MYC and BCL2 rearrangements
* HGBCL, NOS. (6) At least one measurable site of disease (>1.5 cm long axis). (7) No previous treatment for lymphoma. (8) Life expectancy ≥6 months. (9) Left ventricular ejection fraction (LVEF) ≥50% on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO) (10) Patient has adequate liver function:

  * Total bilirubin ≤1.5 x ULN (≤3 x ULN in patients with Gilbert's syndrome).
  * AST (aspartate aminotransferase) and ALT (alanine aminotransferase) ≤3 x ULN.

    o Patients with documented liver involvement: AST and/or ALT ≤5 x ULN. (11) Patient has adequate hematological function, unless due to lymphoma:
  * Hemoglobin ≥9.0 g/dL within 7 days before the first treatment.
  * Absolute neutrophil count of ≥1.0 x 109 cells/L (1,000/μL).
  * Platelet count of ≥75 x 109 cells/L (75,000/μL). Note: Transfusion of RBCs and platelets is allowed to reach the inclusion criteria. In case screening procedures are leading to situations that would exclude the patient from study participation (such as Hb value below entry criteria), the patient may still be enrolled into the trial after consultation with the principal investigator.

    (12) Patient has adequate renal function:
  * Creatinine ≤ 1.5 x ULN, or Creatinine clearance (CrCl) calculated by Cockcroft-Gault formula of ≥ 30 mL/min for patients in whom, in the Investigator's judgment, serum creatinine levels do not adequately reflect renal function.

Exclusion Criteria:

* Patients who meet at least one of the following criteria are not eligible for trial participation:

  1. History of severe cardiac disease: New York Heart Association (NYHA) grade 3-4, congestive heart failure, myocardial infarction or cerebrovascular accident within the past 3 months, unstable arrhythmias, or unstable angina or history of multiple cardiovascular events) or significant pulmonary disease (including obstructive pulmonary disease and history of bronchospasm).

     Note: Congestive heart failure NYHA II patients can be included if they provide an LVEF > 40%.
  2. Patient with current or history of CNS lymphoma.
  3. Patient with uncontrolled severe infection, whether bacterial (e.g., tuberculosis), viral (including, but not limited to severe pneumonia, COVID-19, Epstein-Barr virus [EBV], cytomegalovirus [CMV], hepatitis B, hepatitis C, and HIV], fungal, mycobacterial, or other pathogens (excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics (for IV antibiotics this pertains to completion of last course of antibiotic treatment) within 4 weeks prior to study enrollment.

     Note: Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
  4. Patient with current > Grade 1 peripheral neuropathy.
  5. Any other prior malignancy than non-melanoma skin cancer or stage 0 (in situ) cervical carcinoma, unless treated with curative intent, and without relapse since 2 years, or low grade prostate cancer, not in need of treatment
  6. Psychiatric illness or condition which could interfere with their ability to understand the requirements of the study.
  7. Known hypersensitivity to hamster ovary (CHO) cell products or to any component of the Zuberitamab, polatuzumab vedotin, obinutuzumab, or glofitamab and/or to the contrast agents used in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
CR rate at C4D1 | 9 weeks
  CR rate, defined as the proportion of patients achieving complete remission at Cycle 4 Day 1.

SECONDARY OUTCOMES:
2-yr Progression-free survival (PFS) rate | 2 years follow-up after EOT
  PFS, defined as the time from first treatment to disease progression (PD) or relapse after complete remission (CR) as per Lugano Classification of 2014, or death due to any cause, whichever occurs first. Patients who have not experienced an event at the time of analysis will be censored at the most recent date of disease assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Li, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China